CLINICAL TRIAL: NCT03854045
Title: Team-based Telemedicine
Brief Title: Exploratory Study Providing Telepsychiatry in the Home With a Clinician Present
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Cynthia L. Arfken, PhD, Professor, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MHEF 2018
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Mental Disorder
Keywords: telepsychiatry; telemedicine; home-based care
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Nonequivalent pre-post
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based (Experimental): Clinicians at the FQHC will identify and offer the opportunity to receive telepsychiatry in the home with 2 clinicians present. The patients are not required to agree to the evaluation to receive the services. The services are entered into their EHR but are not eligible for Medicaid reimbursement.
  Interventions: Other: Telepsychiatry
- Clinic-based (Active Comparator): Clinicians at the FQHC will identify and offer the opportunity to receive telepsychiatry in the clinic with 1 clinican present. The patients are not required to agree to the evaluation to receive the services. The services are entered into their EHR and eligible for Medicaid reimbursement.
  Interventions: Other: Telepsychiatry

INTERVENTIONS:
Other: Telepsychiatry — Receive telepsychiatry with clinician obtaining initial data and presenting it to the psychiatrist

SUMMARY:
Telemedicine can expand access to behavioral health services for people who have difficulty traveling to clinics. Travel can be especially challenging for older adults with mobility issues or access to reliable transportation. Assessment in the home can uncover factors impacting patient's physical and behavioral health. The goals of this project to document benefits and barriers to expanding reimbursement for telemedicine to older patient's home as the originating site.

DETAILED DESCRIPTION:
The goal of this project is to document the benefits and barriers to expanding reimbursement for telemedicine to older patient's home as the originating site. The objectives are:

* Develop training module for midlevel clinicians to be ready for dissemination
* Improved patient outcomes measures on satisfaction with care; functioning and symptoms (anxiety, depression, traumatic stress, sleep apnea, alcohol use and problems)
* Reductions in emergency healthcare utilization and medications prescribed as obtained from electronic health record (EHR) at the Federally Qualified Health Center (FQHC) and self-reports
* Summarize activities and barriers, including communication with primary care provider, identification and improvement of home environmental risks, and assistance to support system

This is an observational study of team-based telepsychiatry in the home for one group and team-based psychiatry in the clinic for the comparison group. The initial assessment will include information and informed consent for treatment, biopsychosocial assessment, summary for the psychiatrist, psychiatric evaluation and recommendations (all standard of care). To that the investigators are adding informed consent for program evaluation with 6 month follow-up with information for re-contacting (3 sources, addresses, email-telephone numbers), and brief administration of selected instruments before informed consent for treatment. If an eligible patient does not want to participate in the research study, the patient would still receive services.

Additional telemedicine sessions and/or therapy sessions will be conducted as medically needed in accordance with quality care. At six months (with one month window on either side) the evaluation packet will be re-administered by the clinician if convenient or by the research assistant either in person or by phone.

The sample size was selected to provide robust indicators of barriers to home based assessments. The comparison group was included to provide a context for the findings. It is anticipated that the home group will have greater problems at baseline than the clinic based comparison group but both will show improvements.

ELIGIBILITY:
Inclusion Criteria:

* patient at FQHC
* referred for psychiatric services
* 50 or older

Exclusion Criteria:

* does not speak English

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 | 6 months
  depressiive symptoms

SECONDARY OUTCOMES:
GAD7 | 6 months
  anxiety symptoms
Home checklist | 6 months
  Problems detected in the home

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Arfken, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No